CLINICAL TRIAL: NCT02733237
Title: Oxytocin Effects on the Tolerance of Infidelity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-04
Record Dates: First submitted 2016-03-30; First posted 2016-04-11 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: oxytocin; infidelity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- male oxytocin group (Experimental): male subjects with oxytocin treatment
  Interventions: Drug: oxytocin treatment
- female oxytocin group (Experimental): female subjects with oxytocin treatment
  Interventions: Drug: oxytocin treatment
- male placebo group (Placebo Comparator): male subjects with placebo treatment
  Interventions: Drug: placebo treatment
- female placebo group (Placebo Comparator): female subjects with placebo treatment
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: oxytocin treatment — intranasal administration of oxytocin (40 IU)
  Arms: female oxytocin group; male oxytocin group
Drug: placebo treatment — intranasal administration of placebo (40 IU)
  Arms: female placebo group; male placebo group

SUMMARY:
To investigate whether intranasal oxytocin (40 IU) treatment can influence the tolerance of infidelity in males and females.

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo controlled design, investigators plan to investigate the effect of oxytocin treatment on the tolerance of infidelity. Male and female subjects would firstly see a neutral face of the opposite sex presented with a sentence descried their fidelity or infidelity behavior (sexual or emotional) in a relationship. Next the participant will rate the attractiveness, likability and trustworthiness of each individual, and whether they would like to have a short/long relationship with him/her. After that there will be some implicit attitude tasks to test their implicit attitude towards potential partners exhibiting previous fidelity or and infidelity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* pregnant,menstruating,taking oral contraceptives
* medical or psychiatric illness.

Ages: 19 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
attitude towards fidelity and infidelity of potential mate. | 1 hour
  attitude is measured by the rating scores for likability, attractiveness and trustworthiness

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- China, Sichuan, Chengdu, Sichuan, China